CLINICAL TRIAL: NCT01547325
Title: Double-Blind, Single-Site, Pilot Study of NanoDOX Hydrogel Versus Placebo Hydrogel for Dehisced Surgical Wounds.
Brief Title: Study of NanoDOX Hydrogel vs Placebo for Dehisced Surgical Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NanoSHIFT LLC (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-DOX-NT/005
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Dehisced Surgical Wounds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NanoDOX Hydrogel (Experimental)
  Interventions: Drug: NanoDOX 1% doxycycline monohydrate Hydrogel
- Placebo Hydrogel (Placebo Comparator)
  Interventions: Drug: placebo hydrogel

INTERVENTIONS:
Drug: NanoDOX 1% doxycycline monohydrate Hydrogel — 1% doxycycline monohydrate hydrogel
  Arms: NanoDOX Hydrogel
Drug: placebo hydrogel — placebo hydrogel
  Arms: Placebo Hydrogel

SUMMARY:
The purpose of this study is to determine the effects of NanoDOX Hydrogel versus Placebo Hydrogel on Dehisced Surgical Wounds.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Women of childbearing potential must have a negative urine pregnancy test at screening and at baseline, and:
* Agree to use a double-barrier method of contraception during their participation in this study;

  * condoms (with spermicide) and hormonal contraceptives OR
  * condoms (with spermicide) and intrauterine device OR
  * intrauterine device and hormonal contraceptives OR
  * Abstains from sexual intercourse during their participation in this study OR
  * Is with a same-sex partner and does not participate in bisexual activities where there is a risk of becoming pregnant
* Have a full-thickness dehisced surgical wound that is between 1.2cm2 and 4 cm2 at initial screening
* Be able to apply study drug to their wound, or have a reliable and capable caregiver do it
* Subjects will have adequate blood flow to the wound as defined by transcutaneous oxygen tension (TcpO2) of >30mmHg recorded over intact epidermis at the dehisced surgical wound margin
* Non-infected (Quantitative bacterial count of < 1.0 x 105 cfu)

Exclusion Criteria:

* Less than 18 years of age
* Pregnant or lactating woman or a female of childbearing potential who is not practicing acceptable form of birth control
* Allergic to tetracycline, minocycline, demeclocycline, or any other known tetracycline derivative
* Tested positive for a doxycycline-resistant infection
* Have undergone treatment with system corticosteroid or immunosuppressive therapy in the past 2 months
* Currently undergoing dialysis for renal failure
* Have participated in another clinical research trial within the last 30 days
* Subject has wounds resulting from any cause other than surgical intervention (diabetes, electrical burn, arterial insufficiency, chemical or radiation insult)
* Active or previous (within 60 days prior to the study screening visit) chemotherapy
* Active or previous (within 60 days prior to the study screening visit) radiation to the affected wound area to be treated by investigational drug or placebo
* Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements standard-of-care self-care requirements, and all study-related follow up visit requirements
* History of sickle cell anemia
* History of infection with Human Immunodeficiency Virus
* History of other immunodeficiency disorders
* Severe anemia - Hgb < 10 g/dL (males) or < 9 g/dL (females)
* Severe malnutrition (Albumin < 3.0 gm/dl; > 10% weight loss in preceding 6 weeks)
* Subjects that the Investigators deems unstable and/or require intensive monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The rate of 100% wound closure during the 8-week study | subjects will be followed during their participation in the study for an average of 8 weeks

SECONDARY OUTCOMES:
Safety endpoint | subjects will be followed during their participatoni in the study for an average of 8 weeks
  determined by wound score, area of the wound, and the assessment of wound effluent cytokine, chemokine, protease, and patient reported pain and quality of life questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States